CLINICAL TRIAL: NCT06369532
Title: Stop Worrying, Learn to Let go Through a Combination of Neurostimulation and Psychotherapy
Brief Title: Combination of Neurostimulation and Psychotherapy to Stop Worrying
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONZ-2023-0460
Record Dates: First submitted 2024-01-22; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Active tDCS; Sham tDCS
Keywords: transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be allocated into two groups randomly (using a code). The psychotherapist, the study managers and the patients will not be aware of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS group (Active Comparator): Patients will receive active tDCS during the therapy.
  Interventions: Device: Active tDCS
- Sham tDCS group (Sham Comparator): Patients will receive sham tDCS during the therapy.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — During the whole therapy period, active tDCS group will receive active tDCS after CBT. They also receive active home-based tDCS.
  Arms: Active tDCS group
Device: Sham tDCS — The sham tDCS group will receive sham tDCS after CBT. They also receive sham home-based tDCS.
  Arms: Sham tDCS group

SUMMARY:
This study aims to investigate whether the combination of transcranial Direct Current Stimulation (tDCS) and cognitive-behavioral therapy (CBT) is more effective for treating repetitive negative thinking (RNT) in patients with the symptom of high rumination. High ruminators will be included (Group1, active tDCS-CBT group; Group2, sham tDCS-CBT group). All patients will receive active or sham tDCS.

DETAILED DESCRIPTION:
A psychoeducational CBT-based group intervention called 'Drop It' specifically for the treatment of repetitive negative thinking (RNT), which has been proved to be effective in reducing RNT. tDCS is one of the emerging non-invasive brain stimulations techniques that can also be used to alter RNT. Our aim is to explore the therapeutic effect of this combination.

The study consists of 2 stages. In the first stage the participants will come to the university hospital for 7 weeks CBT sessions (the Drop It intervention), with one session per week. After each CBT session, both groups will receive sham or active tDCS. Stimulation will be applied for 30 min after the CBT session.

In the second stage, after the 7th weekly CBT session, participants will take the devices home to apply daily home-based tDCS stimulations for 4 weeks. After 4 weeks, participants will return to the university hospital for the final CBT session.

Neuroimaging: Electroencephalogram (EEG) and functional Near-Infrared Spectroscopy (fNIRS) scan will be used to measure electrical activity and cortical hemodynamic activity in the brain. Both of these methods are non-invasive neuroimaging techniques which are done by placing electrodes on the scalp to pick up the signals produced by the brain.

EEG and fNIRS scans will be performed at baseline and after 3 months therapy.

To examine the effect of the worry course combined with tDCS on thinking and acting, the investigators will ask the participants to complete various questionnaires that assess the nature and extent of worry, the presence of depressive complaints, the presence of anxiety problems and the extent of quality of life as experienced by the participants. Participants will also be evaluated by a psychiatrist from the service. This evaluation will take place at baseline, just after the end of the Drop It course and after a 3-month follow-up. Two questionnaires will also be used after each session to measure the state rumination following the combination therapy of CBT and tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Generalized anxiety disorder (GAD)
* Depressive disorder

Exclusion Criteria:

* other psychiatric pathology than GAD or depression screened by senior psychiatrist by means of the Mini-International Neuropsychiatric Interview (MINI) and psychiatric anamnesis
* Abuse of alcohol, drugs or medication other than prescribed by general practitioner or psychiatrist
* no consent to participate in measurement (questionnaire, fNIRS or EEG)
* Insufficient knowledge of the current language (Dutch)
* Acute or chronic suicidality
* Acute psychosis or manic depressive disorder
* Inability to commit to 8 sessions of Cognitive-Behavioral Therapy (CBT) or receive 4 weeks of transcranial Direct Current Stimulation (tDCS).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
the therapeutic effect of the combination therapy for repetitive negative thinking | Baseline, up to 7 weeks' therapy and up to 3 months' therapy
  Questionnaires including the Penn State Worry Questionnaire (PSWQ, range 16-80), the Leuven adaptation of the rumination on sadness Scale (LARSS, range 21-105) , and the Ruminative Response Scale (RRS, range 22-88) will be used to measure the alteration of repetitive negative thinking. Higher scores suggest a higher level of worry or rumination. The Beck Depression Inventory (BDI), the Hamilton Depression Rating Scale (HDRS) and other related questionnaires will also be included.
the consolidation effect of tDCS on CBT | up to 7 weeks' therapy and up to 3 months' therapy
  The Self-Critical Rumination scale (SCRS, range 0-40) and the Perseverative Thinking Questionnaire (PTQ, range 0-60) will be measures after each session (8 sessions in total). Higher scores suggest a higher level of self-critical ruminative thoughts or repetitive negative thinking.

SECONDARY OUTCOMES:
Change of neuroimaging data | Baseline and up to 3 months' therapy
  The alteration of brain activity when performing cognitive task measured by EEG and emotional regulation task measured by fNIRS.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Baeken, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baeken C, Wu GR, Rogiers R, Remue J, Lemmens GM, Raedt R. Cognitive behavioral based group psychotherapy focusing on repetitive negative thinking: Decreased uncontrollability of rumination is related to brain perfusion increases in the left dorsolateral prefrontal cortex. J Psychiatr Res. 2021 Apr;136:281-287. doi: 10.1016/j.jpsychires.2021.02.011. Epub 2021 Feb 13. PMID 33621914
- [Result] Sathappan AV, Luber BM, Lisanby SH. The Dynamic Duo: Combining noninvasive brain stimulation with cognitive interventions. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:347-360. doi: 10.1016/j.pnpbp.2018.10.006. Epub 2018 Oct 9. PMID 30312634
- [Result] Dedoncker J, Baeken C, De Raedt R, Vanderhasselt MA. Combined transcranial direct current stimulation and psychological interventions: State of the art and promising perspectives for clinical psychology. Biol Psychol. 2021 Jan;158:107991. doi: 10.1016/j.biopsycho.2020.107991. Epub 2020 Nov 21. PMID 33232800